CLINICAL TRIAL: NCT04697459
Title: Chronic Intradialytic Exercise: a Cardioprotective Role
Brief Title: Chronic Intradialytic Exercise : a Cardioprotective Role
Acronym: EX-CHRODIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-09-14
Record Dates: First submitted 2020-12-14; First posted 2021-01-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Renal Failure
Keywords: exercise; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: * Acute phase : standard HD versus HD with acute intradialytic exercise (in HD-EX group only);
  * Chronic phase : before and after an exercise training program of 16 weeks (HD-EX group) as well as before and after 16 weeks of standard HD (HD group)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD-EX (patient with intradialytic exercise) (Experimental): will be enrolled in a 16 week intradilatytic exercise program.
  Interventions: Other: chronic phase; Other: acute phase
- HD (patients with standard HD) (No Intervention): patients with standard hemodialysis (e.g. without exercise).

INTERVENTIONS:
Other: chronic phase — 1h of intradialytic execise, starting 30 min after hemodialysis beginning : 30 min of low-intensity (Borg Scale 11-14) aerobic exercise + 30 min of resistance training, frequency : 3 times a week for 16 weeks.
  Arms: HD-EX (patient with intradialytic exercise)
Other: acute phase — 30 min of low-intensity (Borg Scale 11-14) aerobic exercise, starting 30 min after hemodialysis beginning
  Arms: HD-EX (patient with intradialytic exercise)

SUMMARY:
The main objective is to assess the effects of chronic intradialytic physical exercise on myocardial remodelling and regional function.

DETAILED DESCRIPTION:
Background: Hemodialysis patients have a mortality rate 50 times higher than in the general population, and the cause remains cardiovascular in more than half of the cases. A deleterious morphological and functional cardiac remodelling is well established in these patients, the causes of which are both the presence of factors specific to renal disease (hemodynamic and non-hemodynamic) and co-morbidities (diabetes, hypertension, etc. .) but also to the hemodialysis (HD) procedure itself, due to the sudden hemodynamic changes it imposes, leading to repeated episodes of intradialytic hypotension (HID) and myocardial stunning. The latter are now documented as direct contributors to the increased mortality observed in HD patients compared to the general population. The introduction of intradialytic physical exercise in the therapeutic program of HD patient is now recommended and practised routinely in many countries, in Scandinavia in particular. Several meta-analyses have clearly established its safety. The beneficial role of chronic intradialytic exercise in improving dialysis efficiency, mental health and quality of life, as well as the inflammatory status of HD patients is also clearly demonstrated. Chronic intradialytic exercise is also associated with improvements in overall fitness level, a parameter closely linked to cardiovascular mortality. Applied acutely during dialysis, it could play a cardioprotective role (e.g; limiting myocardial stunning), allowing haemodynamic and cardiac functional stabilization during HD. However, to our knowledge, no study to date has investigated the long-term effects of intradialytic exercise on remodelling and overall and regional heart function.

Aims: The main objective is to assess the effects of chronic intradialytic physical exercise on myocardial remodelling and regional function. The secondary objectives are to evaluate the effect of acute intradialytic exercise on myocardial stunning as well as the effect of chronic physical exercise on macro and microcirculatory vascular function, inflammation, physical fitness and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* No medical contraindication to physical activity
* Life expectancy greater than 6 months
* Patients on haemodialysis for more than 3 months

Exclusion Criteria:

* Pregnancy

  * Valvular heart disease,
  * Unstable coronary artery disease
  * Arteriopathy obliterating of the lower limbs stage III and IV
  * Musculoskeletal problems
  * Severe respiratory disease
  * BMI> 35
  * Pacemaker, cardiac stimulation and automatic implantable defibrillator
  * Heart transplant
  * Uncontrolled arterial hypertension
  * Ejection fraction <45%

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in myocardial longitudinal deformations | Acute phase : just before and 90 and 210 minutes within standard dialysis or dialysis including acute exercise.
  Myocardial longitudinal linear deformations (in percent) will be assessed by high-resolution echocardiography in deformation imaging mode.
Changes in myocardial longitudinal deformations | Chronic phase : before (week 0) and after (week 17) an exercise training program of 16 weeks; each time in the same conditions as in acute phase (e.g. just before and 90 and 210 minutes within standard dialysis or dialysis including acute exercise).
  Myocardial longitudinal linear deformations (in percent) will be assessed by high-resolution echocardiography in deformation imaging mode.
Changes in myocardial circumferential deformations | Acute phase : just before and 90 and 210 minutes within standard dialysis or dialysis including acute exercise.
  Myocardial circumferential linear deformations (in percent) will be assessed by high-resolution echocardiography in deformation imaging mode.
Changes in myocardial circumferential deformations | Chronic phase : before (week 0) and after (week 17) an exercise training program of 16 weeks; each time in the same conditions as in acute phase (e.g. just before and 90 and 210 minutes within standard dialysis or dialysis including acute exercise).
  Myocardial circumferential linear deformations (in percent) will be assessed by high-resolution echocardiography in deformation imaging mode.
Changes in left ventricular torsion | Acute phase : just before and 90 and 210 minutes within standard dialysis or dialysis including acute exercise.
  Left ventricular torsion (in degree) will be assessed by high-resolution echocardiography in deformation imaging mode.
Changes in left ventricular torsion | Chronic phase : before (week 0) and after (week 17) an exercise training program of 16 weeks; each time in the same conditions as in acute phase (e.g. just before and 90 and 210 minutes within standard dialysis or dialysis including acute exercise).
  Left ventricular torsion (in degree) will be assessed by high-resolution echocardiography in deformation imaging mode.

SECONDARY OUTCOMES:
Changes in arterial rigidity | before (week 0) and after (week 17) an exercise training program of 16 weeks
  Measurement of pulse wave velocity (m/s) by photo-plethysmography at rest before dialysis.
Changes in Physical fitness | before (week 0) and after (week 17) an exercise training program of 16 weeks
  The six-minute walking test (meters); maximal isometric force (newtons) during a knee-extension test and handgrip test using a dynamometer.
Health-related Quality of life | before (week 0) and after (week 17) an exercise training program of 16 weeks
  The 36-Item Short Form Health Survey questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Changes in carotid intimal-media wall thickness | before (week 0) and after (week 17) an exercise training program of 16 weeks
  The intimal plus media wall thickness (mm) of the right carotid artery will be measured using high-resolution echography.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Obert, Pr., Study Chair — Avignon University
Locations (2):
- France (2):
  - Centre Hemodialyse AIDER sante, Nîmes, Gard
  - ATIR, Avignon, Vaucluse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Josse M, Patrier L, Isnard M, Turc-Baron C, Grandperrin A, Nottin S, Mandigout S, Cristol JP, Maufrais C, Obert P. Cardioprotective Effect of Acute Intradialytic Exercise: A Comprehensive Speckle-Tracking Echocardiography Analysis. J Am Soc Nephrol. 2023 Aug 1;34(8):1445-1455. doi: 10.1681/ASN.0000000000000149. Epub 2023 Apr 18. PMID 37071035